CLINICAL TRIAL: NCT02608983
Title: Hydrocolloids as Functional Food Ingredients for Gut Health
Acronym: HYFFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: CyberColloids Ltd. (Industry); University of Reading (Other); The Hebridean Seaweed Company (Industry); Marigot Ltd. (Industry); Industrias Roko, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REC/09/003
Record Dates: First submitted 2015-07-08; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Seaweed; Hydrocolloid; Functional Food; Dietary Fibre; Prebiotic; Low molecular weight polysaccharides; Alginate; Agar; HYFFI; Low molecular weight seaweed derived hydrocolloids as functional food ingredients; subjects
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Experimental)
  Interventions: Dietary Supplement: Agar H1CC2013
- Treatment 2 (Experimental)
  Interventions: Dietary Supplement: Agar H1CC2012
- Treatment 3 (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Agar H1CC2013 — Following a 28-day washout one 250ml drink / day containing 8g of agar H1CC2013 as part of normal diet for 28 days
  Arms: Treatment 1
Dietary Supplement: Agar H1CC2012 — Following a 28-day washout one 250ml drink / day containing 8g of agar H1CC2012 as part of normal diet for 28 days
  Arms: Treatment 2
Dietary Supplement: Maltodextrin — Following a 28-day washout one 250ml drink / day containing 8g of maltodextrin as part of normal diet for 28 days
  Arms: Treatment 3

SUMMARY:
Seaweeds are a natural source of nutrients, and dependent on the variety, are rich in dietary fibre, proteins, essential vitamins and minerals. However this resource is highly underexploited. Countries such as Japan, China, North and South Korea are large consumers of edible seaweed while exposure in Western countries is much lower and mainly as industrially extracted seaweed derivatives, a common additive in many food and healthcare products. Seaweeds have been associated with a number of human gut promoting health benefits such as decreasing faecal transit time through the gastrointestinal tract thus preventing constipation and resulting in a reduced exposure to harmful substances (decreasing colon cancer risk). These health benefits can be attributed to seaweeds high dietary fibre content. Interestingly, the food and healthcare industry already utilize seaweed-extracted fibre in the manufacturing process thus steering the way forward towards the development of novel functional food products. These seaweed-extracted fibres are high molecular weight polysaccharides known as hydrocolloids and are non-digestible by humans, hence classified as dietary fibre.

Traditionally, seaweed derived polysaccharides (hydrocolloids) have been used to provide thickening and gelling functionality to food stuffs and other industrial applications however there is emerging evidence to show that lower molecular weight polysaccharides and oligosaccharides derived from these hydrocolloids can also act as a source of soluble fibre and may have prebiotic activity. Recent developments in Japan and Korea have lead to the commercial availability of products containing low molecular weight seaweed derived fibre. There is also some evidence for the beneficial effects of seaweed derived fibre in other key health areas such as cardiovascular health, cancer, diabetes and obesity. However, relatively little is known about the chemical, physio-chemical and fermentation characteristics of seaweed fibre in the human gut. Some hydrocolloids, notably guar gum (plant source), have also been employed for their health promoting properties in the areas of glucose tolerance and cholesterol lowering. However the use of hydrocolloids as functional food ingredients with health benefits for consumers has been rather limited and has focused more on uses in products for diabetics.

It is particularly in the area of gut health that small and medium-sized enterprises (SMEs) involved in hydrocolloid production and processing, can enter the functional food ingredients market by using innovative processing technology. The total dietary fibre content of seaweed can be as high as 75% of the total dry weight and a high proportion of this is soluble. The fibre component essentially comprises the structural polysaccharides i.e. alginate and fucoidan in brown seaweeds, carrageenan, agar and porphyran in red seaweeds and ulvan in green seaweeds. As these fibres are primarily soluble, they form viscous gels as they pass through the gastrointestinal tract. Some of the fibre is fermented in the lower intestine but in general, soluble and insoluble seaweed fibre tends to pass through the gut without being digested. In its natural form as part of the seaweed plant, this fibre is typically high in molecular weight and passes through the gut too rapidly for the gut microflora to utilize it to any great extent. There is therefore a necessity to develop lower molecular weight forms that are more soluble and can be added at higher concentrations to food products without affecting the sensory properties of the product.

The overall aim of the project is to realize an opportunity to produce low molecular weight polysaccharides (LMWP) from alginate- and agar-bearing seaweeds for applications in food & health. The two effective agar and alginate LMWPs, identified by in vitro studies, will be selected for assessment of prebiotic activity in a feeding trial in human volunteers (Ulster University) as part of an European Union (EU) study. The end points to be assessed will be stimulation of beneficial bacteria (bifidogenic effects), increased short chain fatty acid production, beneficial effects on stool formation, and improvements in gut barrier function. Additionally, benefits of the LMWPs towards blood glucose levels (short term and acute) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age 18-55 years
* Non smoking
* BMI >20 and <35kg/m2

Exclusion criteria

* Smoker
* Pregnant and lactating women
* Vegetarians and vegans
* Lactose intolerant individuals
* Diabetes
* Cardiovascular disease
* Autoimmune/ inflammatory disorders
* History of neoplasm
* Recent acute illness and/or chronic prescribed or self-prescribed use of anti-inflammatory agents (including aspirin)
* Use of broad spectrum antibiotics
* Use of drugs active on gastrointestinal motility or laxatives
* Use of dietary supplements (specifically probiotics or prebiotics)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in faecal bacterial composition | up to 28-day treatment period (six/participant in total)
  Fluorescent in situ hybridisation

SECONDARY OUTCOMES:
Short chain fatty acid concentrations | up to 28-day treatment period (six/participant in total)
  Gas Chromatography
Faecal water barrier function bioactivity | up to 28-day treatment period (six/participant in total)
  Trans-epithelial electrical resistance
Bowel habits | 7 days following each faecal sample provision (six diaries/participant in total)
  Faecal diary
Faecal characteristics | up to 28-day treatment period (six/participant in total)
  Faecal sample type by inspection (Bristol Stool Chart)
Faecal output weight | up to 28-day treatment period (six/participant in total)
  Total faecal output weight
Faecal pH | up to 28-day treatment period (six/participant in total)
  pH meter
Food intake | 4 days prior to each faecal sample provision (six diaries/participant in total)
  Food diary analysed using a Food Composition Database
Acute glycaemic response on subset of volunteers (n=20) | Two days (mornings) following crossover intervention study
  Oral glucose tolerance test following 1.Glucose + Alginate H1CC2012, or 2. Glucose